CLINICAL TRIAL: NCT05090137
Title: Quantifying Interstitial and Intravascular Fluid Accumulation by Ultrasound Following Temporary Suspension of Loop Diuretics in Patients With Heart Failure
Brief Title: Quantifying Congestion by Ultrasound
Acronym: QUEST-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: GN18CA427
Record Dates: First submitted 2021-03-26; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Diuretics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diuretic cessation (Other): Participants will be asked to withhold their diuretic therapy (loop diuretics and mineralocorticoid receptor antagonists) 48 hours prior to visit
  Interventions: Other: Diuretics
- Usual diuretic regimen (Other): Participants will take their usual diuretic regimen prior to study visit. At least one week is required between cross-over visits
  Interventions: Other: Diuretics

INTERVENTIONS:
Other: Diuretics — As per group descriptions

SUMMARY:
The investigators will determine the feasibility of identifying and quantifying changes in interstitial and intravascular congestion by imaging in participants with heart failure. The investigators will either continue or temporarily suspend both loop diuretics and mineralo-corticoid antagonists (MRA) for 48 hours in participants with heart failure that is both stable and mild and compare measurements of interstitial (B-lines) and intra-vascular fluids (IVC and JV diameter and renal venous flow) by ultrasound and, in a subset of participants without contra-indications, by cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure
* Plasma NT-proBNP >125ng/L or BNP >35 ng/l
* Left ventricular ejection fraction (LVEF) <50% on prior imaging test
* Treated routinely with a daily dose of loop diuretic
* Receiving other guideline-indicated therapy for heart failure
* Willing to sign the informed consent form
* Greater than 18 years of age

Exclusion Criteria:

* Chronic Kidney Disease Stage 4 or worse (eGFR <30 mL/min/1.73 m²)
* Atrial fibrillation
* Significant valve disease (investigators opinion)
* Breathlessness or chest pain at rest or minor exertion
* Patients unable to lie flat
* Patients deemed too unstable to miss treatment with diuretics for 48 hours
* Patients taking part in another interventional trial
* Any other concomitant condition that in the opinion of the investigator would not allow a safe participation in the study (ie:-pregnancy, significant frailty)
* Patients unwilling or unable to consent
* For patients willing to undergo MRI; contraindication to MRI including claustrophobia, metalworkers, and intra-orbital or intracranial metal (eg:- stents), and non-MRI compliant device.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Differences in ultrasound markers or congestion following continuation or suspension of diuretics for 48 hours. | at baseline
  Differences in interstitial (B-lines) and intravascular (IVC and JV diameter, and renal venous flow) congestion by ultrasound in patients with heart failure following continuation or suspension of diuretics for 48 hours.

SECONDARY OUTCOMES:
The acute variation in interstitial and intravascular congestion on imaging tests following administration of diuretics. | up to 3 hours
  The acute variation in interstitial (B-lines) and intravascular (inferior vena cava, jugular vein diameter and renal venous flow) congestion on imaging tests following administration of diuretics.
The acute variation in biomarkers of congestion, inflammation and myocardial injury following administration of diuretics. | at 3 hours
  The acute variation in biomarkers of congestion (NT-proBNP), inflammation (HsCRP) and myocardial injury (Troponin) following administration of diuretics.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No